CLINICAL TRIAL: NCT00067483
Title: Pilot Study on the Use of the NASA-NEI Dynamic Light Scattering (DLS) Device in Detecting Lens Changes in the Other Eye of Patients With Pre-Senile Cataracts
Brief Title: Pilot Study: Dynamic Light Scattering Device for Studying Early Changes in Cataract
Status: Completed | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030275; 03-EI-0275
Record Dates: First submitted 2003-08-20; First posted 2003-08-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-12-10

CONDITIONS: Cataract
Keywords: Cataract; Pre-Senile; Dynamic Light Scattering (DLS); Light Scattering; Lens; Cataracts
MeSH Terms: conditions — Cataract

SUMMARY:
This study will use a new dynamic light scattering device (DLS), developed jointly by NASA and the NEI, to study pre-senile cataracts (cataracts that develop in patients 55 years old or less). Cataract is a clouding of the lens that interferes with the passage of light to the retinal, impairing visual acuity. DLS uses a low intensity laser light (similar to that used in supermarket checkouts) to measures lens cloudiness. It detects changes in the human lens at the earliest molecular stages of cataract development, when anti-cataract treatment would be most effective in reversing, delaying or preventing cataract formation.

Patients 55 years of age or younger with cataract may be eligible for this study. Candidates will be screened with the following tests and procedures:

* Medical history and physical examination.
* Eye examination, including measurement of visual acuity (vision chart) and eye pressure; examination of pupils and eye movements; dilation of the pupils for examination of the lens and the back of the eye (retina).
* Cataract photography using a camera with a bright flash to assess the status of the cataract and evaluate future changes.
* Blood drawing if necessary for clinical care.

Participants will have a standard eye examination, as described above, plus DLS testing. For this procedure, the patient sits in front of the DLS device, with the chin placed on a chin rest. He or she fixes on a yellow-green target in the center of the camera lens. When the eye is properly aligned, the measurement is taken and the reddish light on the side of the camera lens turns on for 5 seconds. Measurements are taken on three layers of the lens. The procedure takes less than 30 minutes.

Participants will be followed at the NIH clinic once a month for up to 1 year to follow progression of the cataract. The visits will include a repeat of some of the exams listed above.

DETAILED DESCRIPTION:
Recently, a device has been created to determine molecular interactions that occur in the human lens in vivo and non-invasively, called Dynamic Light Scattering Device (DLS). Preliminary studies have shown its potential in the detection of the earliest changes occurring in cataract, at the stage where anti-cataract treatment would theoretically be most effective in reversing, delaying or preventing cataracts. A new DLS device has been developed by NASA physicist Dr. Rafat Ansari using lower energy lasers, miniaturized and contained within a fiber optic tip, and further developed and tested under an NEI-NASA Inter Agency Agreement. We recently conducted a pilot study to evaluate the usefulness and reproducibility of this instrument for quantitating lens changes, and found good reproducibility. We also determined that a useful parameter is mean particle size. We therefore propose to use the new NEI-NASA DLS device to detect and study, non-invasively and in vivo, the earliest molecular cataractous changes that develop rapidly in the lenses of patients less than 55 years of age, otherwise called pre-senile cataracts.

ELIGIBILITY:
* INCLUSION CRITERIA

Patients 55 years of age or younger with cataracts (pre-senile cataracts) will be admitted to this study.

Ten subjects who have cataracts and who are 55 years of age or younger, of either sex, will be recruited. DLS data will be obtained on the eye with no or little cataract every month for a year or until cataract surgery is required. AREDS grading will be utilized but will not be used as a protocol end point.

EXCLUSION CRITERIA

Patients who have uveitis, glaucoma and who are thought to be at risk for an adverse reaction to pupil dilation, or have a history of allergic reaction to one of the dilating agents that will be used.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15
Dates: Start 2003-08-15; Study Completion 2007-12-10

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - NASA-John Glenn Research Center, Cleveland, Ohio

REFERENCES:
- [Background] Ansari RR, Datiles MB 3rd. Use of dynamic light scattering and Scheimpflug imaging for the early detection of cataracts. Diabetes Technol Ther. 1999 Summer;1(2):159-68. doi: 10.1089/152091599317378. PMID 11475288